CLINICAL TRIAL: NCT00627068
Title: The Role of Nitric Oxide Synthase in Circulating Progenitor Cell Function
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Yerem Yeghiazarians, Assistant Clinical Professor, University of California, San Francisco
Other Study IDs: HL086917
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular; vasodilation; endothelium; Subjects with high cardiovascular risk
MeSH Terms: conditions — Cardiovascular Diseases; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: High cardiovascular risk age over 61 years.
- 2: Low Cardiovascular risk age over 61.
- 3: High cardiovascular risk age over 25 but under 61.
- 4: Low cardiovascular risk age over 25 under 61.

SUMMARY:
Our main hypothesis is that EPC function is impaired in some populations with high cardiovascular risk as a result of reduced eNOS-dependent NO production.

DETAILED DESCRIPTION:
To determine if a correlation exists between EPC function and eNOS-dependent NO production in EPCs from populations with high versus low cardiovascular risk:

1. High and low cardiovascular risk subjects will be identified based on age or history of cardiovascular disease. Endothelial function will be measured by ultrasound.
2. EPCs will be isolated from peripheral blood of these subjects. EPC function will be assessed by measuring adhesion to endothelium, migration, proliferation, and differentiation, and compared to their expression and activity of eNOS.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent and comply with study requirements
* Adult of 18 years or older
* Subjects willing to provide blood and tissue samples

Exclusion Criteria:

* Failure to give informed consent.
* Those unable to consent for themselves.
* Those who cannot read English.
* Patients on Viagra, Levitra, or Cialis
* Patients with malignant disease
* Patients with hematological abnormalities
* Patients with fevers of unknown origin
* Severe comorbidity or alcohol/drug dependence
* Women who are post-menopausal and on hormone replacement therapy, or premenopausal and on birth control pills (premenopausal women will be screened verbally and then by assay of LH and FSH levels in blood samples to identify women in the follicular phase of their menstrual cycle, to reduce variability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population in both low and high risk groups should represent the general population.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yerem Yeghiazarians, M.D, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, Department of Cardiology, San Francisco, California, United States